CLINICAL TRIAL: NCT06615115
Title: Effects of an External and Combined Focus of Attention-Instructed Exercise Program on Postural Stability and Dual-Task Walking in Parkinson's Disease: A Randomized, Assessor-Blinded, Controlled Trial
Brief Title: The Effect of Different Types of Focus Instructions in Parkinson's Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, Assistant Professor, PT, PhD, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LPar24
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; Cognitive Deficit in Attention; Feedback, Psychological; Gait, Festinating
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants who meet the inclusion criteria will be randomized into external focus of attention, combined focus of attention, and control groups. The same exercise program will be administered to all three groups by the same physiotherapist. The exercise program will last for 6 weeks, with sessions held three times a week. Although the exercises will be the same, the instructions given to the patients will vary by group. Assessments will be repeated at the beginning of treatment and at the end of the 6th week by a blinded evaluator.
Who Masked: Outcomes Assessor
Masking Description: The participant will do the evaluations but no info will be given about the randomization adn groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group1: Exercises with External Attention Focus Instructions (Experimental): Throughout the descriped exercise program, the physiotherapist will guide the participants using only external focus of attention instructions.
  Example: Go over the red block. (10 rounds )
  Interventions: Other: Exercise
- Group 2: Exercises with Combined Attention Focus Instructions (Experimental): The exercise program given to the External Focus of Attention group will also be administered to this group. While guiding the exercises, the physiotherapist will use a combination of both external and internal focus of attention instructions to direct the participants.
  Example: Pass over the red block by pulling your knees up as high as you can.
  Interventions: Other: Exercise
- Grup 3: Exercises with no instructions (Control Group) (Experimental): The same exercise program given to the other groups will also be administered to this group but no instruction will be given to this group.
  Example: Take 10 turn around the track, passing over the blocks
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — All participants will perform a total body stretching exercise for 10 minutes, followed by 10 minutes of obstacle course navigation, 10 minutes of balance training (including tandem walking, balance board exercises, single-leg balance, and two-legged reaching exercises), and will conclude with 10 minutes of strength training exercises.

SUMMARY:
Parkinson's disease is the most common progressive neurodegenerative movement disorder. Common movement impairments in Parkinson's include balance and walking difficulties. These impairments lead to falls, increased levels of functional dependency, and a decrease in quality of life. Exercise in Parkinson's patients improves their functional symptoms in daily life, enhancing both motor and non-motor skills, and consequently increases their quality of life. Recently, various additional methods have been developed to increase the effectiveness of exercise in Parkinson's rehabilitation and to contribute to motor skills. Focus of attention instructions are fundamental concepts in motor function learning. External focus of attention has been shown to facilitate motor function development, reduce postural instability, and improve dual-task walking by being easier to remember. In Parkinson's patients who experience freezing phenomena, internal focus of attention instructions enhance walking stability and movement control, thereby reducing the risk of falls. However, there are no studies on the combined focus of attention instructions in Parkinson's patients. This study is designed as a randomized controlled, single-blind, prospective trial to examine the effects of a combination of internal and external focus of attention instructions on walking, balance parameters, quality of life, and patient satisfaction levels, taking into account the presence of freezing phenomena in Parkinson's patients.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the most common progressive neurodegenerative movement disorder. Common movement impairments in Parkinson's include balance and walking difficulties. These impairments lead to falls, increased levels of functional dependency, and a decrease in quality of life. Such deficits are associated with the acquisition of motor function skills. Although PD patients are open to learning, they experience challenges with motor planning. Therefore, individuals with PD may require additional training, sensory input, and motor education for the permanence and ease of motor skill acquisition.

The difficulties PD patients face with complex commands indicate that they can learn in a feedforward manner, but they show inconsistencies in the use of automatic functions. This inconsistency results in challenges in adapting to variable situations and performing complex activities (like balance and walking). Exercise in Parkinson's patients improves their functional symptoms in daily life, enhancing both motor and non-motor skills, and consequently increasing their quality of life. Recently, various additional methods have been developed to enhance the effectiveness of exercise in Parkinson's rehabilitation and to contribute to motor skills. One commonly used method to address deficits in motor behavior is motor learning activities, which involve repetitive movements and ensure continuity.

Many studies have shown that the concept of focus of attention contributes to the efficiency and learning of various motor functions, particularly balance. Individuals with Parkinson's are highly receptive to external stimuli, so a focus-based strategy during balance and walking training can improve these skills. Focus of attention instructions are fundamental concepts in motor function learning. External focus of attention facilitates motor function development, reduces postural instability, and improves dual-task walking. In Parkinson's patients who experience freezing phenomena, internal focus of attention instructions enhance walking stability and movement control, thereby reducing the risk of falls. However, there are no studies on the combined focus of attention instructions in Parkinson's patients.

This study is designed as a randomized controlled, single-blind, prospective trial to examine the effects of a combination of internal and external focus of attention instructions on walking, balance parameters, quality of life, and patient satisfaction levels, considering the presence of freezing phenomena in Parkinson's patients. Approximately 48 individuals with Parkinson's disease without freezing phenomena will participate in an exercise program for six weeks, three days a week. Participants will be randomized into a combined focus group, an external focus group, and a control group. Assessments will be repeated at the beginning and end of the six-week exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn and Yahr Stage II or III
* Individuals between the ages of 50 and 70 who can walk independently but have balance disorders
* Having a score between 21-56 on the Berg Balance Scale
* Having a score between 24-30 on the Mini Mental State Test
* Having agreed to participate in the study (Not having a freezing phenomenon)
* Being in the Medication-on period

Exclusion Criteria:

* Having malignancy and metabolic diseases
* Having had Cerebrovascular Accident before
* Other neurological disease history
* Presence of cognitive problems
* Presence of visual or hearing disorders
* Presence of deep brain pacemaker
* Presence of freezing phenomenon (persons with Freezing of Gait Questionnaire FOG-Q above zero)
* Presence of dyskinesia

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | baseline, six weeks after the baseline
  This is a 14-item scale that measures the ability to maintain balance during dynamic tasks. It is rated on a scale of 0 to 4 points, with a maximum total score of 56. As the total score decreases, the risk of falling increases.
  0 to 20 points: Indicates that the individual is dependent on a wheelchair and has a 100% risk of falling. 21 to 40 points: Suggests that the individual has a moderate risk of falling and may be able to walk with assistance. 41 to 56 points: Indicates that the individual can ambulate independently with a low risk of falling.
Time Up and Go Dual Task | baseline, six weeks after the baseline
  The test assesses balance, walking, and functionality during activities. The TUG-Dual Task evaluates walking abilities and attention management by asking participants to solve a simple math problem or perform another cognitive task while walking. Patients will be assessed for functionality, walking speeds, and balance evaluations. If the duration lasts more than 12 seconds, there is a risk of falling.

SECONDARY OUTCOMES:
The Parkinson's Disease Questionnaire-39 (PDQ-39) | baseline, six weeks after the baseline
  The PDQ-39 is a PD specific health status questionnaire comprising 39 items. Respondents are requested to affirm one of five ordered response categories according to how often, due to their PD, they have experienced the problem defined by each item. Items are grouped into eight scales that are scored by expressing summed item scores as a percentage score ranging between 0 and 100 (100¼more health problems).

OTHER OUTCOMES:
Likert Scale Questionnaire | baseline, six weeks after the baseline
  Likert scale is a measurement tool that combines multiple Likert-type questions. It is defined as the creation of two or more Likert-type questions to address a single research problem, and using the average values of these questions during the analysis phase. The aim is to determine individuals' average attitudes on these topics based on the combined values of all questions. To determine the scope of the patient's treatment, 5 questions and a high score of 10 are evaluated. The highest score is 50, indicating that the person is satisfied with the treatment; as the score decreases, satisfaction with the treatment decreases.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Koçak, PT, Principal Investigator — Bahcesehir University, Faculty of Health Sciences, Department of Physiotherapy; Pelin Pişirici, PT, PhD, Study Director — Bahcesehir University, Faculty of Health Sciences
Locations (1):
- Atafiz Tıp Merkezi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No